CLINICAL TRIAL: NCT02560103
Title: An Observational Study to Investigate the Effects of Rapid Travel
Brief Title: An Observational Study to Investigate the Effects of Rapid Transmeridian Travel
Status: Completed | Type: Observational
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: VP-VEC-162-0101
Record Dates: First submitted 2015-09-21; First posted 2015-09-25 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Jet Lag Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single group: No treatment
  Interventions: Other: Transmeridian travel across multiple time zones

INTERVENTIONS:
Other: Transmeridian travel across multiple time zones

SUMMARY:
Observational study to investigate circadian rhythm patterns

ELIGIBILITY:
Inclusion Criteria:

* Ability and acceptance to provide written consent
* Men or women between 18-75 years
* Body Mass Index of ≥ 18 and ≤ 30 kg/m2

Exclusion Criteria:

* History (within the 12 months prior to screening) of psychiatric disorders
* Major surgery, trauma, illness or immobile for 3 or more days within the past month
* Pregnancy or recent pregnancy (within 6 weeks)
* A positive test for drugs of abuse at the screening visit
* Any other sound medical reason as determined by the clinical investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2015-09; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Effects of transmeridian travel on nighttime sleep after transmeridian travel measured by Polysomnography (PSG) | 4 days
Karolinska Sleepiness Scale (KSS) in subjects who experienced rapid transmeridian travel. | 4 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Santa Monica Clinical Trials, Santa Monica, California
  - The Center for Sleep & Wake Disorders, Chevy Chase, Maryland